CLINICAL TRIAL: NCT00714883
Title: A Prospective, Multi-Center Study of the Conor Cobalt Chromium Reservoir Based Stent (NevoTM) With Sirolimus Elution in Native Coronary Artery Lesions (NEVO RES-II)
Brief Title: Conor Cobalt Chromium Reservoir Based Stent With Sirolimus Elution in Native Coronary Artery Lesions
Acronym: NEVO RES-II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The NEVO™ stent will not be commercialized. Cordis decided to close the study after 3 years. This decision took the absence of safety signals into account.
Sponsor: Cordis US Corp. (Industry)
Collaborators: Conor Medsystems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-07
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Disease
Keywords: drug-eluting stents; Percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: NEVO™ Sirolimus-eluting Coronary Stent System — Intervention will consist of percutaneous coronary intervention for treatment of lesions in native coronary arteries using standard coronary intervention techniques. Intervention will include treatment with the NEVO™ Sirolimus-eluting Coronary Stent System.
  Other Names: NEVO

SUMMARY:
The primary objective of this study is to evaluate the target lesion failure rate of the NEVO Sirolimus-eluting Coronary Stent System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with atherosclerotic CAD ;
* The subject must be >/= 18 years of age;
* Female of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment;
* Diagnosis of angina pectoris as defined by stable angina pectoris Canadian Cardiovascular Society Classification (Class I, II, III) OR non-ST segment elevation acute coronary syndrome (Braunwald Classification B&C) OR OR non-ST segment elevation myocardial infarction ≥ 48 hours from the time of study index procedure OR asymptomatic subjects with a positive stress test;
* Indicated treatment of up to two lesions in one or two major coronary arteries (1 target lesion in each of 2 vessels or 2 target lesions in 1 vessel). The target vessel diameter must be >/= 2.25mm and </= 3.5 in diameter (visual estimate);
* Target lesion length </= 28 mm able to be treated with a single stent. If required, additional Conor Sirolimus stents should be used to treat dissections, etc
* Patient or Legally Authorized Representative must provide written informed consent prior to the procedure using a form that is approved by the Independent Ethics Committee.
* The patient is willing to comply with all specified follow-up evaluations.
* The target lesion has been successfully crossed with the intracoronary guidewire which is positioned intraluminally in the distal vessel.
* The target lesion diameter stenosis is >50% and <100% based on a visual estimate.

Exclusion Criteria:

* ST-elevation MI within 72 hours prior to the index procedure and/or creatine kinase (CK) >2 times the local laboratory upper limits of normal on the day of the index procedure.
* The patient has undergone target vessel revascularization within 6 months prior to the intended enrolment procedure.
* Prior stent within 5 mm of target lesion(s);
* Ostial target lesion(s);
* Unprotected left main coronary disease with >/= 50% stenosis;
* Angiographic evidence of thrombus within target lesion(s);
* Total coronary occlusion or TIMI grade 0 or 1 in the target vessel;
* Bifurcation disease involving a side branch >/= 2 mm in diameter;
* Target lesion(s) within a coronary bypass graft (e.g., saphenous vein or arterial graft);
* Significant calcification or angulation in the target vessel that, in the Investigator's opinion, may preclude stent delivery and deployment;
* Recipient of heart transplant;
* Subject with a life expectancy less than 12 months;
* Known allergies to the following: aspirin, any thienopyridine, heparin, cobalt chromium, contrast agent (that cannot be managed medically), or sirolimus that cannot be managed medically;
* The patient has contraindication to ASA or to any thienopyridine agent.
* Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the study endpoints;
* Known bleeding or hypercoagulable disorder;
* Known or suspected active infection at the time of the study procedures;
* Subject is known to be a prisoner, mentally incompetent, and/or alcohol or drug abuser;
* Subject has had major surgical or interventional procedures unrelated to this study within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study, or planned coronary PCI through the end of the study.
* The patient is currently taking systemic immunosuppressant therapy;
* The patient has co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
target lesion failure (TLF) | 12 months post procedure

SECONDARY OUTCOMES:
Lesion success | Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrejs Erglis, MD, Principal Investigator — P. Stradina Clinical-University Hospital; Prof. Bruno Scheller, Principal Investigator — Klinik für Innere Medizin III, Universitätsklinikum des Saarlandes
Locations (2):
- Klinik für Innere Medizin III, Universitätsklinikum des Saarlandes, Homburg/Saar, Germany
- P. Stradina Clinical - University Hospital, Riga, Latvia

REFERENCES:
- [Derived] Otake H, Honda Y, Courtney BK, Shimohama T, Ako J, Waseda K, Macours N, Rogers C, Popma JJ, Abizaid A, Ormiston JA, Spaulding C, Cohen SA, Fitzgerald PJ. Intravascular ultrasound results from the NEVO ResElution-I trial: a randomized, blinded comparison of sirolimus-eluting NEVO stents with paclitaxel-eluting TAXUS Liberte stents in de novo native coronary artery lesions. Circ Cardiovasc Interv. 2011 Apr 1;4(2):146-54. doi: 10.1161/CIRCINTERVENTIONS.110.957175. Epub 2011 Mar 8. PMID 21386089